CLINICAL TRIAL: NCT06299319
Title: Evaluating the Feasibility, Clinical Effects, and Safety of Psilocybin-assisted Psychotherapy for Treatment-resistant Obsessive-compulsive Disorder: An Open-label Clinical Trial
Brief Title: Feasibility, Clinical Effects, and Safety of Psilocybin-assisted Psychotherapy for Treatment-resistant OCD
Acronym: PAP-OCD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 149-2021
Record Dates: First submitted 2024-02-15; First posted 2024-03-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: psilocybin; psychedelics; obsessive-compulsive disorder; clinical trial
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Psilocybin 25 mg (Experimental): Participants will receive a 25 mg dose of psilocybin, twice throughout the trial, with two weeks in between doses.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — The psilocybin used in this study meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of psilocybin. The psilocybin will be administered twice during the trial, in conjunction with supportive therapy.
  Other Names: PEX010

SUMMARY:
Psilocybin, the chemical component of "magic mushrooms", has been administered with psychotherapy in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects. There is interest to see if similar effects may be provided in those with obsessive compulsive disorder (OCD).

The purpose of this study is to evaluate the safety, feasibility, and clinical effects of psilocybin administration in those with OCD. Ten participants with treatment-resistant OCD will receive two doses of 25mg of psilocybin under supportive conditions, two weeks apart. The investigators hypothesize that two sessions of psilocybin 25mg administered under supportive conditions to participants with treatment-resistant OCD will lead to significant reductions in OCD symptoms.

DETAILED DESCRIPTION:
Literature suggests that up to 40 percent of individuals with OCD do not respond to conventional treatment and experience treatment resistant OCD (TROCD) (1, 2). Psilocybin, the chemical component of "magic mushrooms", has been administered with psychotherapy in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects (3). Results of these trials have led to growing calls for transition to clinical use, as well as increased research for other mental health disorders. It is presumed that psilocybin's therapeutic effects are induced by the psychedelic "trip", which is dependent on serotonin 2A receptor (5-HT2AR) activation (4, 5). All studies have used psilocybin in conjunction with psychotherapy involving two therapists present during full-day dosing sessions. There is a need for more data in the TROCD population as there is only one clinical trial published for this specific population, followed by various case reports.

Using a proof-of-concept, open-label, clinical trial approach, 10 participants with TROCD will receive 2 doses of 25mg of psilocybin, with two weeks between each dosing day. The objectives of this study are as follows:

1. To assess the safety, and feasibility, of psilocybin, administered with psychological support to adult participants with TROCD. Hypothesis 1: The investigators will be able to recruit and retain ten participants with TROCD for the duration of the trial and that psychedelic-assisted psychotherapy for obsessive compulsive disorder (PAP-OCD) will be safe in those with TROCD, as measured by monitoring adverse events and using the Columbia Suicide Severity Rating Scale (C-SSRS).
2. To assess the clinical effects of PAP in those with TROCD. Hypothesis 2: Two sessions of psilocybin (25mg) administered under supportive conditions to participants with TROCD will lead to significant reductions in OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) when comparing baseline to Week 3.
3. Provide pilot data on the effect of psilocybin and supportive therapy on TROCD in preparation of a future larger RCT.

Overview of Study Design:

All 10 participants will follow the same study design. Each participant will undergo a screening assessment where they will complete lab tests, and clinical and psychiatric assessments to determine eligibility. Following the screening visit, participants will undergo a washout period where they will be tapered off concomitant medications over a medication the participant is being tapered off (based on the half-life of the medication) and the participant's preference for the length of the tapering period. All medications will require a minimum of a 2-week tapering period with the exception of fluoxetine which will require a minimum of 4-weeks. Additional time may be added at the discretion of the study investigator. During this period, there will be weekly check-ins with the study physician.

At study Visit 2 (Baseline, V2), participants will complete a series of questionnaires and assessments, preparatory therapy with trained study therapists, and undergo a brain functional magnetic resonance imaging (fMRI). The preparatory therapy sessions will build a therapeutic alliance, and provide psychoeducation about, and set intentions for, the psilocybin session. To reduce participant burden, baseline can be broken up into multiple days, however all assessments must be completed within 7-days of the first dose. At study Visit 3 (V3), neurophysiological measurements will be performed.

Upon completion of V2 and V3, participants will undergo the first psilocybin dosing session at Visit 4 (V4) where they will receive an active dose (25mg) of psilocybin in conjunction with supportive therapy. The psilocybin session will last 5 to 6 hours and will be conducted in the existing psychedelic treatment suite developed at the Centre for Addiction and Mental Health (CAMH). Two trained study therapists will be supporting each participant during the dosing session. After 5 hours of dose administration, participants will be evaluated for safety by the study psychiatrist and discharged home in the company of a caregiver or a family member.

On the day after the dosing session (Visit 5, V5) and one-week after the dosing session (Visit 6, V6), participants will be asked to complete the same questionnaires that were done at Baseline (V2) and will undergo an integrative therapy session with the trained study therapist. At Visit 7 (V7), 2-weeks after the first psilocybin dose, participants will undergo the second psilocybin dosing session where they will receive an active dose (25mg) of psilocybin in conjunction with supportive therapy.

On the day after the second dosing session (Visit 8, V8) and one-week after the second dosing session [3-weeks after dose 1] (Visit 10, V10), participants will be asked to complete the same questionnaires that were done at Baseline (V2) and will undergo an integrative therapy session with the trained study therapist. Between Visit 8 (V8) and Visit 10 (V10), during study Visit 9 (V9), the same neurophysiological measurements will be performed as during Visit 3 (V3). Follow-up assessments will also occur at 6, 9, and 12 weeks (Visit 11, 12, and 13) after the second psilocybin dosing session. The same questionnaires administered at Baseline (V2) will be repeated at each of these study visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years old;
* Are outpatients
* Must be deemed to have capacity to provide informed consent;
* Must sign and date the informed consent form;
* Stated willingness to comply with all study procedures;
* Ability to read and communicate in English, such that their literacy and comprehension is sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent;
* Primary The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of obsessive compulsive disorder (OCD) based on medical records and assessment using the Structured Clinical Interview for DSM-5 (SCID-5) administered at the first screening visit;
* Participants diagnosed with treatment-resistant OCD defined as individuals with a score of ≥ 16 on the YBOCS (i.e. moderate symptom severity) and that have not responded to two or more separate pharmacological interventions and one or more trials of cognitive behavioural therapy (CBT); there is no upper limit on the number of treatment failures;
* Individuals with an estimated glomerular filtration rate (eGFR) above 40mL/min/1.73m2 and all blood work within normal limits as assessed by clinical laboratory tests at Screening (V1)
* Ability to take oral medication;
* Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation;
* Individuals who are willing to and have tapered off current OCD medications for a minimum of 2-weeks prior to Baseline (V2) and whose physician confirms that it is safe for them to do so;
* Individuals who are willing to and have tapered off current inhibitors of 5'-diphospho-glucuronosyltransferase (UGT)1A9 and 1A10, aldehyde dehydrogenase inhibitors (ALDHs) and alcohol dehydrogenase inhibitors (ADHs) for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and for the duration of the study and whose physician confirms that it is safe for them to do so; and
* Agreement to adhere to Lifestyle Considerations (section 4.5) throughout study duration.

Exclusion Criteria:

* Pregnant as assessed by a urine pregnancy test at Screening (V1) and Baseline (V2) or individuals that intend to become pregnant during the study or are breastfeeding;
* Treatment with another investigational drug or other intervention within 30 days of Screening (V1);
* Have initiated psychotherapy in the preceding 12 weeks prior to Screening (V1);
* Have a DSM-5 diagnosis of substance use disorder (use of tobacco and prescribed opioids are permitted) within the preceding 6 months;
* Have active suicidal ideation as determined by the C-SSRS and/or clinical interview. Significant suicide risk is defined by suicidal ideation as endorsed by items 4 or 5 of the C-SSRS;
* Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder; psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history and the SCID-5 clinical interview;
* Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I or II disorder as determined by the family medical history form and discussions with the participant;
* Have contraindications to transcranial magnetic stimulation (TMS) as determined by the transcranial magnetic stimulation adult safety screen (TASS) questionnaire;
* Have a history of seizures;
* Are taking anticonvulsants or benzodiazepines (Lorazepam up to 2mg/day is acceptable);
* Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment;
* Use of classic psychedelic drugs within the previous 12 months; OR
* Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of administering psilocybin (25 mg) in adults with treatment-resistant OCD | Screening Period, Intervention (2 weeks), Follow-up after 2nd dosing session (up to 10 weeks after 2nd dose)
  Percentage of participants recruited and retained
Incidence of adverse events (Safety and Tolerability) | Screening Period, Intervention (2 weeks), Follow-up after 2nd dosing session (up to 10 weeks after 2nd dose)
  Frequency of dropouts attributed to adverse effects or serious adverse events
Change in the Yale-Brown Obsessive-Compulsive Scale (YBOCS) total score from baseline | Baseline (Day -1) to Week 3 (Day 21)
  The Yale-Brown Obsessive-Compulsive Scale is a test to rate the severity of obsessive-compulsive disorder symptoms. It is a 10-item scale, with questions 1-5 regarding obsessions, and questions 6-10 regarding compulsions. Each item is scored from 1-4, for a total possible score of 40.
  Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Proportion of participants who respond to treatment | Baseline (Day -1) to Week 3 (Day 21)
  Response to treatment defined as a 35 percent or more reduction of the Yale-Brown Obsessive-Compulsive Scale (YBOCS) total score, and remission defined as a score of less than or equal to 7 on the YBOCS.
  The Yale-Brown Obsessive-Compulsive Scale is a test to rate the severity of obsessive-compulsive disorder symptoms. It is a 10-item scale, with questions 1-5 regarding obsessions, and questions 6-10 regarding compulsions. Each item is scored from 1-4, for a total possible score of 40.
  Higher scores represent a more severe condition.
Changes in Patient Health Questionnaire (PHQ-9) from Baseline to Week 3 | Baseline (Day -1) to Week 3 (Day 21)
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  It is a 9-item scale, with each item score ranging from 0 ("Not at all") to 3 ("Nearly every day") for a total possible score of 27.
  Higher scores represent a more severe condition.
Change in the Clinical Global Impression (CGI) scale from Baseline to Week 3 | Baseline (Day -1) to Week 3 (Day 21)
  The Clinical Global Impression (CGI) scale is a 3-item observer-rated scale that measures illness severity, global improvement or change, and therapeutic response. The "Severity" and "Global Improvement or Change" items are scored on a 7-point scale, ranging from 0-7. The "Therapeutic Response" item is scored from 1-16.
  Higher scores represent a worse outcome.
Change in the World Health Organization Quality of Life Short Version (WHOQOL-BREF) score from Baseline to Week 3 | Baseline (Day -1) to Week 3 (Day 21)
  The World Health Organization Quality of Life Short Version (WHOQOL-BREF) is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains quality of life and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5.
  Higher scores represent worse quality of life.
Change in World Health Organization Disability Assessment Schedule (WHODAS 2.0) from Baseline to Week 3 | Baseline (Day -1) to Week 3 (Day 21)
  WHODAS 2.0 is an instrument that assesses functioning. The instrument produces domain-specific scores for six different functioning domains - cognition, mobility, self-care, getting along, life activities (household and work) and participation.
Change in Generalized Anxiety Disorder (GAD-7) scores from Baseline to Week 3 | Baseline (Day -1) to Week 3 (Day 21)
  The GAD-7 measures severity of anxiety symptoms. It is a 7-item scale, with each item ranging from 0 ("Not at all") to 3 ("Nearly every day"), for a total possible score of 21.
  Higher scores represent a more severe condition.
Changes in behavioural assessments for well-being (Warwick-Edinburgh Mental Wellbeing Scale; WEMWBS) from Baseline to Week 3 | Baseline (Day -1) to Week 3 (Day 21)
  WEMWBS is a scale which has been validated for the measurement of mental wellbeing. It is a 14-item scale consisting of positively worded statements, ranging from 1 ("None of the time") to 5 ("All of the time").
  Higher scores represent greater wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Gwyneth Zai, MD, MSc, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch MH, Landeros-Weisenberger A, Kelmendi B, Coric V, Bracken MB, Leckman JF. A systematic review: antipsychotic augmentation with treatment refractory obsessive-compulsive disorder. Mol Psychiatry. 2006 Jul;11(7):622-32. doi: 10.1038/sj.mp.4001823. Epub 2006 Apr 4. PMID 16585942
- [Background] Pallanti S, Quercioli L. Treatment-refractory obsessive-compulsive disorder: methodological issues, operational definitions and therapeutic lines. Prog Neuropsychopharmacol Biol Psychiatry. 2006 May;30(3):400-12. doi: 10.1016/j.pnpbp.2005.11.028. Epub 2006 Feb 28. PMID 16503369
- [Background] Perkins D, Sarris J, Rossell S, Bonomo Y, Forbes D, Davey C, Hoyer D, Loo C, Murray G, Hood S, Schubert V, Galvao-Coelho NL, O'Donnell M, Carter O, Liknaitzky P, Williams M, Siskind D, Penington D, Berk M, Castle D. Medicinal psychedelics for mental health and addiction: Advancing research of an emerging paradigm. Aust N Z J Psychiatry. 2021 Dec;55(12):1127-1133. doi: 10.1177/0004867421998785. Epub 2021 Mar 21. PMID 33745287
- [Background] Halberstadt AL, Koedood L, Powell SB, Geyer MA. Differential contributions of serotonin receptors to the behavioral effects of indoleamine hallucinogens in mice. J Psychopharmacol. 2011 Nov;25(11):1548-61. doi: 10.1177/0269881110388326. Epub 2010 Dec 8. PMID 21148021
- [Background] Madsen MK, Fisher PM, Burmester D, Dyssegaard A, Stenbaek DS, Kristiansen S, Johansen SS, Lehel S, Linnet K, Svarer C, Erritzoe D, Ozenne B, Knudsen GM. Psychedelic effects of psilocybin correlate with serotonin 2A receptor occupancy and plasma psilocin levels. Neuropsychopharmacology. 2019 Jun;44(7):1328-1334. doi: 10.1038/s41386-019-0324-9. Epub 2019 Jan 26. PMID 30685771

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT06299319/Prot_SAP_000.pdf